CLINICAL TRIAL: NCT04416620
Title: The Impact of a Pharmaceutical Care Model on Improving Polycystic Ovary Syndrome Associated Factors Amongst Females in Jordan and Syria
Brief Title: The Impact of a Pharmaceutical Care Model on Improving Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-PHA 2
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Anxiety; Depression; QOL; Biochemical parameters; Lifestyle modifications; pharmacist; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants in the active group received the usual care delivered at the community pharmacies at both countries plus the pharmaceutical care service designed by the research group and provided by the clinical pharmacist, an experienced female with extensive knowledge on PCOS. The intervention was delivered via oral advice and recommendations, and written material, with a special focus on diet and exercise. Participants in the control group received the usual care only and did not receive the pharmaceutical care service.
  Following the intervention, both groups were followed up for four months and re-interviewed at the community pharmacy.
Who Masked: Participant
Masking Description: The study is a single-blinded randomized controlled trial. The patients 'study groups were only known for the clinical pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The active group of Syria (Active Comparator): Participants in the active group received the 'pharmacist standard counseling' plus the 'pharmaceutical care service' designed by the research group. Both services were delivered by one female clinical pharmacist who has a Master's degree in pharmaceutical sciences, 5-year work experience in community pharmacies, and comprehensive knowledge of PCOS. The time it took to deliver the counseling and education to each participant in the active group was formally assessed. This time assessment excluded data collection and questionnaire filling time (which was planned to take around 15 min).
  Participants in the active group received the usual care delivered at the community pharmacies plus the pharmaceutical care service designed by the research group and provided by the clinical pharmacist. The intervention was delivered via oral advice and recommendations, and written material, with a special focus on diet and exercise.
  Interventions: Other: The PCOS pharmaceutical care service
- The control group of Syria (No Intervention): Participants in the control group received the usual care only which is the 'pharmacist standard counseling' involved dispensing the prescribed medication (delivered by the pharmacist in charge), counseling on how to take the dispensed medications, and a brief reply to questions if asked by the participants. The 'pharmacist standard counseling' followed what was normally delivered to females with PCOS by pharmacists working at community pharmacies in both countries. This 'pharmacist standard counseling' was established based on what was observed and reported by the project research team after viewing the usual pharmacists' interaction with females with PCOS for two weeks in each country before the start of the study.
  Participants in the control group were informed that the educational intervention (the pharmaceutical care service) will be delivered to them after the end of the study (for ethical reasons).
- The active group of Jordan (Active Comparator): Participants in the active group received the usual care delivered at the community pharmacies plus the pharmaceutical care service designed by the research group and provided by the clinical pharmacist. The intervention was delivered via oral advice and recommendations, and written material, with a special focus on diet and exercise.
  Interventions: Other: The PCOS pharmaceutical care service
- The control group of Jordan (No Intervention): Participants in the control group received the usual care only which is the 'pharmacist standard counseling' involved dispensing the prescribed medication (delivered by the pharmacist in charge), counseling on how to take the dispensed medications, and a brief reply to questions if asked by the participants. The 'pharmacist standard counseling' followed what was normally delivered to females with PCOS by pharmacists working at community pharmacies in both countries. This 'pharmacist standard counseling' was established based on what was observed and reported by the project research team after viewing the usual pharmacists' interaction with females with PCOS for two weeks in each country before the start of the study.
  Participants in the control group were informed that the educational intervention (the pharmaceutical care service) will be delivered to them after the end of the study (for ethical reasons).

INTERVENTIONS:
Other: The PCOS pharmaceutical care service — The intervention was provided in the format of oral plus written information. The information provided included the importance of exercise and motivational messages to exercise more at home or in the gym.
  The 2nd part was about the importance of decreasing the stress levels. Participants were informed to perform a simple breathing exercise on daily basis twice a day.
  The 3rd part aimed at improving participants' diets. They were informed to follow specific diet recommendations and to avoid certain types of food, explaining to them how it may negatively affect their PCOS condition.
  The 4th part was about the PCOS treatment that was discussed with the participants. Females were advised on the importance of using their correct treatment. They were informed of the importance of adhering to their prescribed medications, accepting that it was a long-term treatment plan, and to consult with their specialist if their treatment was not effective, or in the case of medication side effects.
  Arms: The active group of Jordan; The active group of Syria

SUMMARY:
The primary aim of this study was to estimate the prevalence of anxiety disorder and depression amongst Syrian and Jordanian women who are suffering from PCOS in Damascus and Amman.

The secondary aim was to assess the effectiveness of a PCOS pharmaceutical care service on selected patient's biochemical parameters, QOL, anxiety, and depression scale. The third aim is to identify the factors associated with QOL, anxiety and depression scores' change across the study.

Null Hypothesis (research hypothesis):

The intervention of PCOS pharmaceutical care service will lead to no significant differences in patient's depression, anxiety, QOL, and some biochemical parameters in comparison to females who will not receive this intervention in both Syria and Jordan.

Alternative Hypothesis (research hypothesis):

The intervention of PCOS pharmaceutical care service will have a significant impact on patient's depression, anxiety, QOL, and some biochemical parameters in comparison to patients who will not receive this intervention in both Syria and Jordan.

DETAILED DESCRIPTION:
The information provided in the PCOS pharmaceutical care service was delivered in the format of oral plus written information (most important facts to remember and take-home messages regarding lifestyle modifications). The information provided included the importance of exercise and motivational messages to exercise more at home or in the gym. Participants were informed of previous study results which showed that 8-12 weeks of exercise can ameliorate cardiovascular risk factors and improve mental health.

The second part of the educational service was about the importance of decreasing the stress levels. The participants were informed that markers of oxidative stress were found to be out of range in PCOS women and that it was proven beneficial to do breathing exercises to reduce stress. It was clarified that the breathing exercise does not only relieve stress but also may help to gain better sleep and relieve anxiety symptoms. Participants were informed to perform a simple breathing exercise on daily basis (twice a day, morning and night) where they inhale through the nose for the account of four, and then exhale through the nose for the count of four, with the possibility to increase the counting to 6 then to 8.

The third part of the educational service aimed at improving participants' diets. They were informed to follow specific diet recommendations as follows:

to consume the majority of their daily calories prior to 12 pm (shown to improve insulin and glucose levels and decrease testosterone levels), to focus on food with low glycemic load e.g. chicken, meat, eggs and avocado (shown to decrease insulin levels).

to increase their vitamin C and calcium intake e.g. kiwi, orange and lemons (shown to improve body mass index and menstrual abnormalities, along with other PCOS-related symptoms).

to include adequate magnesium intake in their diet e.g. legume, spinach, broccoli, banana and pineapple (shown to lower the risk of heart disease, diabetes, and stroke).

to increase chromium intake, found in onions, garlic, grapefruit and tomatoes (shown to help regulate insulin and glucose levels).

to increase their consumption of omega-3, found in food such as tuna, salmon, fish, and walnuts (shown to help in decreasing androgen levels and testosterone).

In addition, participants were informed to avoid or to minimize certain types of food, explaining to them how it may negatively affect their PCOS condition. Such food types included caffeine beverages (as it may increase the estrogen level and affect fertility).

hydrogenated oils including margarine, corn oil, and coffee creamers (as it decreases the HDL (the good cholesterol), and increases the LDL (the bad cholesterol).

white sugary foods like cookies, cakes, and candies (as it can increase glucose levels).

dairy products (since it can cause allergic reactions and digestion problems, in addition to raising the testosterone levels).

Processed food (because it has a negative effect on insulin level). PCOS treatment was also discussed (orally only) with the participants (Fourth part of the service). Females were advised on the importance of using their correct treatment, for example using the pill for hormonal balance. They were informed of the importance of adhering to their prescribed medications, accepting that it was a long term treatment plan, and to consult with their specialist if their treatment was not effective, or in the case of medication side effects.

ELIGIBILITY:
Inclusion Criteria:

* Females who had a doctor-diagnosis of PCOS.
* Above the age of 16.
* Able to complete the 4-month study.

Exclusion Criteria:

* Females with an old diagnosis of PCOS with no doctor visit in the past month.
* Can not speak and understand Arabic.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females.
Enrollment: 118 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety prevalence | At baseline
  Anxiety prevalence assessment using the Beck Anxiety Inventory. The BAI scale, consisted of 21-multiple-choice questions, with 4-point scale indicating the degree of anxiety severity (0-3; all questions were scored positively). Points were summed to produce a total measure score, indicating four levels of anxiety severity: 0-7 reflecting minimal level of anxiety, 8-15 reflecting mild level of anxiety, 16-25 reflecting moderate level of anxiety and 26-63 reflecting severe level of anxiety. The possible score for each participant ranged from 0 to 63. Lower scores indicated better anxiety symptoms.
Depression prevalence | At baseline
  Depression prevalence assessment using the Beck Depression Inventory. The BDI is a 4-point scale (0-3) indicating the level of depression severity, with the score referring to six levels: 0-10 indicating the ups and downs reported by the participant were normal, 11-16 reflecting mild mood disturbances, 17-20 reflecting borderline clinical depression, 21-30 reflecting moderate depression, 31-40 reflecting severe depression, and over 40 reflecting extreme depression. The possible score for each participant ranged from 0 to 63. The BDI Questionnaire evaluates pessimistic attitude, loss of appetite, sad mood and feelings of guilt. Lower scores indicated better depression symptoms.
Anxiety scale | Change from Baseline and follow-up (up to 17 weeks)
  Levels of Anxiety severity and mean score assessment were done by the Beck Anxiety Inventory.
  The BAI scale, consisted of 21-multiple-choice questions, with 4-point scale indicating the degree of anxiety severity (0-3; all questions were scored positively). Points were summed to produce a total measure score, indicating four levels of anxiety severity: 0-7 reflecting minimal level of anxiety, 8-15 reflecting mild level of anxiety, 16-25 reflecting moderate level of anxiety and 26-63 reflecting severe level of anxiety. The possible score for each participant ranged from 0 to 63. Lower scores indicated better anxiety symptoms.
Depression scale | Change from Baseline and follow-up (up to 17 weeks)
  Levels of Depression severity and mean score assessment were done by the Beck Depression Inventory.
  The BDI is a 4-point scale (0-3) indicating the level of depression severity, with the score referring to six levels: 0-10 indicating the ups and downs reported by the participant were normal, 11-16 reflecting mild mood disturbances, 17-20 reflecting borderline clinical depression, 21-30 reflecting moderate depression, 31-40 reflecting severe depression, and over 40 reflecting extreme depression. The possible score for each participant ranged from 0 to 63. The BDI Questionnaire evaluates pessimistic attitude, loss of appetite, sad mood and feelings of guilt. Lower scores indicated better depression symptoms.
Quality of Life scale assessment | Change from Baseline Quality of Life and follow-up (up to 17 weeks)
  Quality of Life assessment using the polycystic ovary syndrome health-related QOL questionnaire (PCOSQ).
  It has a 30 questions about symptoms related to menstruation and mood. It can identify seven factors affecting the QOL in PCOS women including: emotional disturbance, hirsutism, weight concerns, infertility, menstrual symptoms, menstrual predictability and acne. The QOL was analyzed individually as a continuous scale out of seven to assess the QOL in patients (the higher the score is, the better the QOL is). After that, each question of the 30 questions included in the PCOSQ questionnaire was analyzed, and the mean score within each question was obtained and compared between baseline and follow-up. After that, each domain included in the QOL questionnaire was analyzed individually. Mean score of each domain was obtained and compared between baseline and follow-u to assess the impact of lifestyle modifications on that domain.
Blood pressure assessment | Change from Baseline Blood Pressure and follow-up (up to 17 weeks)
  Systolic and diastolic blood pressure measurements were measured using the right arm, twice after a 10-min rest and averaged by using the gold standard, mercury sphygmomanometers
Blood Glucose levels | Change from Baseline Blood Glucose levels and Follow-up (up to 17 weeks)
  Blood Glucose levels assessment using the Multi-parametric device.
Blood Cholesterol levels | Change from Baseline Blood Cholesterol levels and follow-up (up to 17 weeks)
  Blood Cholesterol levels assessment using the Multi-parametric device.
Blood Triglycerides levels | Change from Baseline Blood Triglycerides levels and Follow-up (up to 17 weeks)
  Blood Triglycerides levels assessment using the Multi-parametric device.
Body Mass Index | Change from Baseline Body mass index and Follow-up (up to 16 weeks)
  the Body Mass Index was calculated for each participant depending on their weight and hight.

SECONDARY OUTCOMES:
Smoking frequency | Change from Baseline Smoking frequency and Follow-up (up to 17 weeks)
  smokers participants recorded the number of cigarettes smoked per day.
Hooka frequency | change from Baseline Hooka frequency and Follow-up (up to 17 weeks)
  the frequency hooka habits was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Iman A Basheti, Phd, Principal Investigator — ASU; Kinda T Alkoudsi, Master's, Principal Investigator — ASU
Locations (4):
- Five branches of Pharmacy 1, Amman, Jordan
- Syria (3):
  - Almazra pharmacy, Damascus
  - Alwafaa pharmacy, Damascus
  - Kinda Pharmacy, Damascus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benson S, Hahn S, Tan S, Mann K, Janssen OE, Schedlowski M, Elsenbruch S. Prevalence and implications of anxiety in polycystic ovary syndrome: results of an internet-based survey in Germany. Hum Reprod. 2009 Jun;24(6):1446-51. doi: 10.1093/humrep/dep031. Epub 2009 Feb 16. PMID 19223290
- [Result] Laggari V, Diareme S, Christogiorgos S, Deligeoroglou E, Christopoulos P, Tsiantis J, Creatsas G. Anxiety and depression in adolescents with polycystic ovary syndrome and Mayer-Rokitansky-Kuster-Hauser syndrome. J Psychosom Obstet Gynaecol. 2009 Jun;30(2):83-8. doi: 10.1080/01674820802546204. PMID 19533486
- [Result] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291
- [Result] Thomson RL, Buckley JD, Lim SS, Noakes M, Clifton PM, Norman RJ, Brinkworth GD. Lifestyle management improves quality of life and depression in overweight and obese women with polycystic ovary syndrome. Fertil Steril. 2010 Oct;94(5):1812-6. doi: 10.1016/j.fertnstert.2009.11.001. Epub 2009 Dec 11. PMID 20004371
- [Result] Vigorito C, Giallauria F, Palomba S, Cascella T, Manguso F, Lucci R, De Lorenzo A, Tafuri D, Lombardi G, Colao A, Orio F. Beneficial effects of a three-month structured exercise training program on cardiopulmonary functional capacity in young women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Apr;92(4):1379-84. doi: 10.1210/jc.2006-2794. Epub 2007 Jan 30. PMID 17264174